CLINICAL TRIAL: NCT07046442
Title: Effect of Pulmonary Rehabilitation and Physical Activity on the Symptoms of Long COVID. A Pilot Study
Brief Title: Effect of Pulmonary Rehabilitation and Physical Activity on Long COVID (PuReCOVID)
Acronym: PuReCOVID
Status: Active, not recruiting | Type: Observational
Sponsor: University of Parma (Other)
Collaborators: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Sponsor
Other Study IDs: 28421
Record Dates: First submitted 2025-06-27; First posted 2025-07-01 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Long COVID-19 Syndrome
Keywords: long COVID, Pulmonary rehabilitation, ACBT
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 6 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- A group of patients affected by Long Covid 19 disease
  Interventions: Other: Pulmonary Rehabilitation

INTERVENTIONS:
Other: Pulmonary Rehabilitation — The Active Cycle of Breathing Technique (ACBT), is a structured method aimed at restoring normal breathing patterns, improving respiratory muscle efficiency, and reducing airway irritation.

SUMMARY:
This single-center, observational, longitudinal, retrospective and prospective study investigates the impact of Active Cycle of Breathing Technique (ACBT) and moderate daily physical activity on symptoms associated with long COVID, such as cough, dyspnea, and fatigue. The study aims to assess whether these interventions can moderately alleviate or resolve these symptoms and evaluate their potential association with small airway dysfunction (SAD), as measured by Impulse Oscillometry (IOS).

We will recruit 40 adult patients with long COVID who meet specific inclusion criteria. Participants will perform ACBT twice daily and complete at least 6000 steps per day for six weeks. We will track clinical and lung function parameters, including spirometry, IOS, and exercise capacity.

DETAILED DESCRIPTION:
Long COVID affects approximately 10% of COVID-19 survivors, with symptoms persisting beyond the acute phase and impacting multiple organ systems. While some individuals experience mild to moderate illness, others develop severe complications, such as Acute Respiratory Distress Syndrome (ARDS), increasing the risk of long-term pulmonary dysfunction. There is no universally accepted definition of long COVID, but it is often categorized based on symptom duration: post-acute COVID-19 (symptoms persisting beyond three weeks) and chronic COVID-19 (lasting beyond 12 weeks). According to NICE and the Italian National Institute of Health (ISS), long COVID includes symptoms lasting between 4 and 12 weeks (ongoing symptomatic COVID-19) or beyond 12 weeks (post-COVID-19 syndrome), provided they are not attributable to alternative diagnoses.

Common symptoms include fatigue, dyspnea, cough, and chest pain. Some patients recover spontaneously with rest, symptomatic treatment, and gradual physical activity, while others require targeted rehabilitation. Since 80% of breathing effort relies on the diaphragm, long COVID patients often exhibit altered breathing patterns, such as shallow breathing and increased reliance on accessory muscles, leading to dyspnea, fatigue, and inefficient respiration.

Rehabilitation programs have been shown to improve ambulation, hospital discharge rates, and overall recovery in COVID-19 patients, highlighting their potential role in long COVID management. Pulmonary rehabilitation, particularly the Active Cycle of Breathing Technique (ACBT), is a structured method aimed at restoring normal breathing patterns, improving respiratory muscle efficiency, and reducing airway irritation. ACBT consists of controlled breathing, thoracic expansion exercises, forced expiration, and huffing, facilitating airway clearance and optimizing lung function. Given the association between physical inactivity and worse COVID-19 outcomes, rehabilitation strategies incorporating breathing exercises and physical activity may be beneficial.

Pulmonary function studies indicate that Forced Expiratory Volume in 1 second (FEV1) and the FEV1/FVC ratio generally remain within normal limits after COVID-19 recovery, regardless of disease severity. However, impairments in Mid-Expiratory Flow (MEF25-75%) suggest small airway dysfunction (SAD), which appears independent of disease severity but may contribute to persistent respiratory symptoms. Early detection of pulmonary abnormalities is crucial, and Impulse Oscillometry (IOS) is recommended for assessing SAD. Studies indicate that up to 70-90% of symptomatic long COVID patients exhibit persistent SAD up to five months post-infection, emphasizing the need for ongoing lung function monitoring.

This retrospective and prospective study aims to evaluate whether ACBT, combined with moderate daily physical activity, can alleviate symptoms such as cough, dyspnea, and fatigue in long COVID patients. Effectiveness will be assessed using validated clinical scales, including the Leicester Cough Questionnaire (LCQ), the Modified Medical Research Council (mMRC) dyspnea scale, and the Visual Analog Scale (VAS) for fatigue. Additionally, the study will investigate whether respiratory symptoms correlate with SAD, assessed through IOS by analyzing changes in distal airway resistance (R5-R20) and reactance (X5) before and after a six-week rehabilitation period. The rehabilitation protocol involves performing ACBT twice daily at home for six weeks. Clinical and respiratory functional parameters will be assessed before and after the intervention of six weeks. To ensure adherence, patients will receive instructional materials, including video tutorials and augmented reality tools. Additionally, participants will be encouraged to engage in moderate physical activity, aiming for at least 6,000 steps per day, tracked via smartphone applications.

Participants will be monitored over six weeks, with two scheduled visits: an initial baseline assessment (V1) and a follow-up evaluation (V2).

The study protocol was approved by Ethics Committee in the session of 05/07/2022 with protocol. No. 28421 of 07/06/2021.

Data will be collected in a dedicated electronic Clinical Records Form (CRF). The database will be saved on a password-protected company Personal Computer (PC) which will be updated at each visit and used exclusively for scientific research purposes. At the time of enrollment, each patient will receive an alphanumeric code so that any information collected during the study, and in particular sensitive data, is treated in an anonymous manner. Data reporting patients' identifications will only be used to file patients and collect informed consent.

ELIGIBILITY:
Inclusion Criteria:

* Male or female adults aged ≥18 years;
* Signed informed consent;
* Patients with long COVID
* Patients with or without ventilatory deficit (FEV1/FVC>/≤70% and FVC>/≤80%)
* Patients reporting at least one of the following symptoms: cough, dyspnea, and fatigue at 24 weeks post-infection

Exclusion Criteria:

* Patients with other coexisting chronic lung diseases (asthma, fibrosis, bronchiectasis, sarcoidosis, interstitial diseases, pulmonary hypertension)
* Active smoking patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population will consist of 40 adult patients, referred at outpatient clinic of the Respiratory Disease Unit of the University Hospital of Parma (Italy)
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2022-04-05 (Actual); Primary Completion 2025-02-04 (Actual); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
To investigate whether ACBT and moderate daily physical activity can improve cough (LCQ), dyspnea (mMRC) and fatigue (VAS) associated to Long COVID. | six weeks
  Improvement of cough (LCQ), dyspnea (mMRC) and fatigue (VAS) associated to Long COVID after six weeks of pulmonary rehabilitation

SECONDARY OUTCOMES:
To determine whether respiratory symptoms are associated with small airway dysfunction due to mechanical insult from SARS-CoV infection | six weeks
  Improvement of parameters of the small airways in terms of both distal resistance (R5-R20) and reactance (X5) as assessed by pulse oscillometry (IOS) before and after ACBT.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Parma, Parma, Italy, Italy

IPD SHARING:
Plan to Share IPD: Yes
Data will be collected in a dedicated electronic Clinical Records Form (CRF). The database will be saved on a password- protected company personal computer which will be updated at each visit and used exclusively for scientific research purposes. At the time of enrolment, each patient will receive an alphanumeric code so that any information collected during the study, and in particular sensitive data, will be treated in an anonymous manner. Data reporting patients' identifications will only be used to file patients and collect informed consent.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available during the course of the study. The Investigator will keep paper and electronic copies of all documentation at the Center for a period of at least 7 years after the completion of the study and then he will arrange for its destruction.
Access Criteria: Only the personal delegated to collaborate with this study will be able to access to the database using a password to login.

REFERENCES:
- [Background] Rogliani P, Ora J, Girolami A, Rossi I, de Guido I, Facciolo F, Cazzola M, Calzetta L. Ceiling effect of beclomethasone/formoterol/glycopyrronium triple fixed-dose combination in COPD: A translational bench-to-bedside study. Pulm Pharmacol Ther. 2021 Aug;69:102050. doi: 10.1016/j.pupt.2021.102050. Epub 2021 Jun 12. PMID 34129945
- [Background] Calzetta L, Aiello M, Frizzelli A, Bertorelli G, Chetta A. Small airways in asthma: from bench-to-bedside. Minerva Med. 2022 Feb;113(1):79-93. doi: 10.23736/S0026-4806.21.07268-2. Epub 2021 Jan 26. PMID 33496163
- [Background] Li LY, Yan TS, Yang J, Li YQ, Fu LX, Lan L, Liang BM, Wang MY, Luo FM. Impulse oscillometry for detection of small airway dysfunction in subjects with chronic respiratory symptoms and preserved pulmonary function. Respir Res. 2021 Feb 24;22(1):68. doi: 10.1186/s12931-021-01662-7. PMID 33627138
- [Background] EQ-5D. Accessed January 13, 2022. https://euroqol.org/
- [Background] Ward N. The Leicester Cough Questionnaire. J Physiother. 2016 Jan;62(1):53. doi: 10.1016/j.jphys.2015.05.011. Epub 2015 Aug 29. No abstract available. PMID 26320841
- [Background] Birring SS, Prudon B, Carr AJ, Singh SJ, Morgan MD, Pavord ID. Development of a symptom specific health status measure for patients with chronic cough: Leicester Cough Questionnaire (LCQ). Thorax. 2003 Apr;58(4):339-43. doi: 10.1136/thorax.58.4.339. PMID 12668799
- [Background] Bestall JC, Paul EA, Garrod R, Garnham R, Jones PW, Wedzicha JA. Usefulness of the Medical Research Council (MRC) dyspnoea scale as a measure of disability in patients with chronic obstructive pulmonary disease. Thorax. 1999 Jul;54(7):581-6. doi: 10.1136/thx.54.7.581. PMID 10377201
- [Background] Huskisson EC. Measurement of pain. Lancet. 1974 Nov 9;2(7889):1127-31. doi: 10.1016/s0140-6736(74)90884-8. No abstract available. PMID 4139420
- [Background] Aoyagi Y, Shephard RJ. Habitual physical activity and health in the elderly: the Nakanojo Study. Geriatr Gerontol Int. 2010 Jul;10 Suppl 1:S236-43. doi: 10.1111/j.1447-0594.2010.00589.x. PMID 20590838
- [Background] Tudor-Locke C, Bassett DR Jr. How many steps/day are enough? Preliminary pedometer indices for public health. Sports Med. 2004;34(1):1-8. doi: 10.2165/00007256-200434010-00001. PMID 14715035
- [Background] The Active Cycle of Breathing Techniques, available at https://www.acprc.org.uk/Data/Publication_Downloads/GL-05ACBT.pdf. Assoc Chart Physiother Respir Care. Published online 2011. Accessed January 13, 2022. www.brit-thoracic.org.uk/clinical-information/physiotherapy/physiotherapy-guideline.aspx
- [Background] Lewis LK, Williams MT, Olds TS. The active cycle of breathing technique: a systematic review and meta-analysis. Respir Med. 2012 Feb;106(2):155-72. doi: 10.1016/j.rmed.2011.10.014. Epub 2011 Nov 18. PMID 22100537
- [Background] Kellett C, Mullan J. Breathing control techniques in the management of asthma. Physiotherapy. 2002:88,12; 751-758
- [Background] Sallis R, Young DR, Tartof SY, Sallis JF, Sall J, Li Q, Smith GN, Cohen DA. Physical inactivity is associated with a higher risk for severe COVID-19 outcomes: a study in 48 440 adult patients. Br J Sports Med. 2021 Oct;55(19):1099-1105. doi: 10.1136/bjsports-2021-104080. Epub 2021 Apr 13. PMID 33849909
- [Background] Meeting the challenge of long COVID. Nat Med. 2020 Dec;26(12):1803. doi: 10.1038/s41591-020-01177-6. No abstract available. PMID 33288947
- [Background] Huang C, Huang L, Wang Y, Li X, Ren L, Gu X, Kang L, Guo L, Liu M, Zhou X, Luo J, Huang Z, Tu S, Zhao Y, Chen L, Xu D, Li Y, Li C, Peng L, Li Y, Xie W, Cui D, Shang L, Fan G, Xu J, Wang G, Wang Y, Zhong J, Wang C, Wang J, Zhang D, Cao B. 6-month consequences of COVID-19 in patients discharged from hospital: a cohort study. Lancet. 2021 Jan 16;397(10270):220-232. doi: 10.1016/S0140-6736(20)32656-8. Epub 2021 Jan 8. PMID 33428867
- [Background] Interim guidance on Long-COVID Management Principles. ISS COVID-19 Report no. 15/2021 https://www.iss.it
- [Background] COVID-19 rapid guideline: managing COVID-19. NICE guideline Last updated: 13 April 2022.
- [Background] Gupta N, Sachdev A, Gupta D. Oscillometry-A reasonable option to monitor lung functions in the era of COVID-19 pandemic. Pediatr Pulmonol. 2021 Jan;56(1):14-15. doi: 10.1002/ppul.25121. Epub 2020 Oct 26. No abstract available. PMID 33104290
- [Background] Lopes AJ, Litrento PF, Provenzano BC, Carneiro AS, Monnerat LB, da Cal MS, Ghetti ATA, Mafort TT. Small airway dysfunction on impulse oscillometry and pathological signs on lung ultrasound are frequent in post-COVID-19 patients with persistent respiratory symptoms. PLoS One. 2021 Nov 29;16(11):e0260679. doi: 10.1371/journal.pone.0260679. eCollection 2021. PMID 34843598
- [Background] Lv D, Chen X, Wang X, Mao L, Sun J, Wu G, Lin Z, Lin R, Yu J, Wu X, Jiang Y. Pulmonary function of patients with 2019 novel coronavirus induced-pneumonia: a retrospective cohort study. Ann Palliat Med. 2020 Sep;9(5):3447-3452. doi: 10.21037/apm-20-1688. PMID 33065795
- [Background] Jiandani MP, Salagre SB, Kazi S, Iyer S, Patil P, Khot WY, Patil E, Sopariwala M. Preliminary Observations and Experiences of Physiotherapy Practice in Acute Care Setup of COVID 19: A Retrospective Observational Study. J Assoc Physicians India. 2020 Oct;68(10):18-24. PMID 32978920
- [Background] Barker-Davies RM, O'Sullivan O, Senaratne KPP, Baker P, Cranley M, Dharm-Datta S, Ellis H, Goodall D, Gough M, Lewis S, Norman J, Papadopoulou T, Roscoe D, Sherwood D, Turner P, Walker T, Mistlin A, Phillip R, Nicol AM, Bennett AN, Bahadur S. The Stanford Hall consensus statement for post-COVID-19 rehabilitation. Br J Sports Med. 2020 Aug;54(16):949-959. doi: 10.1136/bjsports-2020-102596. Epub 2020 May 31. PMID 32475821
- [Background] Greenhalgh T, Knight M, A'Court C, Buxton M, Husain L. Management of post-acute covid-19 in primary care. BMJ. 2020 Aug 11;370:m3026. doi: 10.1136/bmj.m3026. No abstract available. PMID 32784198